CLINICAL TRIAL: NCT02821455
Title: Does the End-tidal Concentration Estimate the Blood Concentration of Inhalational Anaesthetics During One-lung Ventilation?
Brief Title: Estimating Blood Concentrations of Anaesthetics During One-Lung Ventilation (OLV)
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Other Study IDs: AC16081
Record Dates: First submitted 2016-06-29; First posted 2016-07-01 (Estimated); Results first posted 2018-08-02 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2017-10

CONDITIONS: One-Lung Ventilation
Keywords: Isoflurane; Sevoflurane; Bispectral Index; Pulmonary Surgical Procedures
MeSH Terms: interventions — Pulmonary Surgical Procedures; One-Lung Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 2 10mL whole blood samples per patient
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lung Surgery with One-Lung Ventilation: A single cohort of patients undergoing one-lung ventilation during lung surgery
  Interventions: Procedure: Lung Surgery with One-Lung Ventilation

INTERVENTIONS:
Procedure: Lung Surgery with One-Lung Ventilation — A single cohort of patients undergoing one-lung ventilation during lung surgery

SUMMARY:
The aims of the study is to determine if end-tidal concentrations of the anaesthetic gases isoflurane and sevoflurane as measured by a standard gas monitor are related to the blood levels during one-lung ventilation.

DETAILED DESCRIPTION:
Measurement of the anaesthetic gases such as isoflurane and sevoflurane allow anaesthetists to gauge their blood levels and in turn their brain levels and so help assess how deep the patient is under anaesthesia. These measurements, made as the patient breathes out, are known as end-tidal concentrations of anesthetic gases and are routinely made with gas monitors. Measurement of blood levels of anaesthetic gases is possible but infrequently done as it is time-consuming, expensive, and requires a scientist in a laboratory with specialized equipment. Depth of anaesthesia is assessed using clinical signs along with end-tidal concentrations though more recently it can be assessed by monitoring the brain's electrical waves. This technique remains controversial.

Mechanically supporting the patient's breathing using only one of the two lungs, known as one-lung ventilation, is used in lung surgery to allow the surgeon to gain access to one side of the chest whilst the anaesthetist supports the lung on the other side. One-lung ventilation markedly alters the exchange of gases in the lungs, including anaesthetic gases. Because of this derangement, it is not known if the end-tidal concentrations are related to blood levels of anaesthetic gases during this type of mechanical ventilation. The aims of the study is to determine if end-tidal concentrations of anaesthetics as measured by a standard gas monitor are related to the blood levels of the gases isoflurane and sevoflurane during one-lung ventilation.

Patients over 18 years old undergoing planned lung surgery with one-lung ventilation and anaesthesia with isoflurane or sevoflurane, and who have a routine tube inserted into an artery in their wrist to monitor blood pressure will be recruited for the study. During the study, two blood samples the size of two teaspoons each will be taken from the tube in the artery and two end-tidal concentration recordings.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18
* Admitted for elective thoracic surgery using one-lung ventilation obtained by the use of a double-lumen endotracheal tube or bronchial blocker.
* Elective surgery planned between 1 August and 30 November 2016
* Planned insertion of an arterial cannula by anaesthetist for routine monitoring of systemic arterial pressure
* Planned inhalational anaesthesia technique with isoflurane or sevoflurane.
* Patients who have provided consent to take part in the study

Exclusion Criteria:

* Patients under the age of 18
* History of malignant hyperthermia
* Emergency thoracic surgery
* Patients who have not consented to take part in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled to undergo elective lung surgery with planned one-lung ventilation, identified from the operative list of a university hospital
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2016-08; Primary Completion 2016-11 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R P Alston, MBChB,FRCA, Principal Investigator — University of Edinburgh
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lung Surgery With One-Lung Ventilation
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lung Surgery With One-Lung Ventilation
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.2 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Correlation Between Blood and End-tidal Isoflurane or Sevoflurane Concentration During One-lung Ventilation
Description: The significance of the correlation between blood and end-tidal isoflurane or sevoflurane concentration during one-lung ventilation
Time Frame: 10 minutes after start of one-lung ventilation
Measure: Number; unit: Correlation coefficient
Arm/Group | Lung Surgery With One-Lung Ventilation
Number analyzed (Participants) | 19
Correlation coefficient | 0.0807

2. Secondary Outcome: Correlation Between Bispectral Index (BIS) and End-tidal Isoflurane or Sevoflurane Concentration During One-lung Ventilation.
Description: The significance of the correlation between BIS and end-tidal isoflurane or sevoflurane concentration during one-lung ventilation.
Time Frame: 10 minutes after start of one-lung ventilation
Population: Data not collected due to insufficient use of Bispectral Index Monitors and temperature monitors by anaesthetists responsible for the study participants at the study site.
Arm/Group | Lung Surgery With One-Lung Ventilation
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Lung Surgery With One-Lung Ventilation
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No